CLINICAL TRIAL: NCT03959774
Title: Assessment of Outpatient Digital Follow-up of Patients Over 70 Years of Age Undergoing Chemotherapy Treatment
Acronym: E-SN@P PROJECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-SN@P PROJECT-IPC 2017-029
Record Dates: First submitted 2019-05-21; First posted 2019-05-22 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer
Keywords: Elderly population; digital monitoring
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- breast or colorectal or lung cancer, age 70 or older (Experimental): breast or colorectal or lung cancer, age 70 or older
  Interventions: Device: IPC NET

INTERVENTIONS:
Device: IPC NET — a digital pack with connected bracelet and connected balance will be given to the patient. IPC NET and Nokia Health applications will be downloaded. Pairing between connected objects and the smartphone will be done during the inclusion visit

SUMMARY:
adherence of digital follow-up in a population of elderly patients.

DETAILED DESCRIPTION:
The use of digital self-questionnaires adapted to elderly patients but also to BrC and Bac could detect the toxicities of chemotherapy and we formulate the hypothesis that the continuous monitoring of these different variables in elderly patients treated with chemotherapy is possible and acceptable to this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years,
2. Patient with an indication of adjuvant chemotherapy showing:

   * Breast cancer
   * Colorectal cancer
   * lung cancer

4. WHO ≤ 3 (WHO index - World Health Organization) 5. Estimated life expectancy> 6 months 6. patients with a smartphone or tablet with an internet connection. It can also be offered to patients whose primary caregiver or the person of trust (including the partner) has a smartphone, an internet connection or a tablet provided that he or she is present more than three times during the week. during chemotherapy to ensure smooth weekly data transfer and filling of questionnaires 7. Signed consent to participation 8. Affiliation to, or beneficiary of, a social security scheme

Exclusion Criteria:

1. Person in emergency situation, person of legal age subject to a legal protection measure (major under guardianship, guardianship or court order), or unable to express his / her consent
2. Impossibility of submitting to the medical examination of the test for geographical, social or psychological reasons
3. Contraindications to the procedure of the study: patient or caregiver living with a patient who does not have a smartphone with an internet connection (patient or caregiver living with a patient)
4. Concurrent participation in another clinical trial
5. Patient unable to understand the quality of life survey and Patient Reported Outcome

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
demonstrate that the adherence rate of digital follow-up is greater than 70% in a population of elderly patients. | 12 months after the last chemotherapy received by the patient
  numerical follow-up compliance rate, defined as the rate of patients who observed the following three rules during the entire course of adjuvant chemotherapy: a minimum weight per week, the wearing of the bracelet for three consecutive days per week, and the weekly response to the digital self-questionnaire. Failure to comply with at least one of these rules will be considered a failure.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tassy, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (4):
- France (4):
  - Institut Sainte Catherine, Avignon
  - CHI des Alpes du Sud, Gap
  - Institut Paoli-Calmettes, Marseille
  - CHU Nice, Nice

IPD SHARING:
Plan to Share IPD: No